CLINICAL TRIAL: NCT01944865
Title: Effect of Intermittent Versus Interval Training on Mountain Bike Cross-country Performance: a Parallel-group Randomized Trial
Brief Title: Interval Training and Performance in Mountain Bikers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Gama Filho (Other)
Responsible Party: Principal Investigator, Tony Meireles dos Santos, Ph.D., Universidade Gama Filho
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: UGF
Record Dates: First submitted 2013-08-31; First posted 2013-09-18 (Estimated); Last update posted 2013-09-18 (Estimated); Status verified 2013-09

CONDITIONS: Physical Activity
Keywords: Aerobic Interval Training; Supramaximal Training
MeSH Terms: conditions — Motor Activity | interventions — High-Intensity Interval Training

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Interval Training (Experimental): The INTV consisted of 7 to 10 repetitions of 4-6 min at the highest intensity sustainable, and in the last 30 s of each repetition was performed a maximal sprint, the active recovery was 4-6 min in intensity from 10 to 15 of scale of perceived exertion CR100.
  Interventions: Other: Interval Training
- Intermittent Training (Experimental): The riders completed 8 to 12 repetitions of 30 s all-out with 4 min of active recovery (10-15 on the CR100 scale).
  Interventions: Other: Intermittent Training

INTERVENTIONS:
Other: Interval Training — The interval training group consisted of 7 to 10 repetitions of 4-6 min at the highest intensity sustainable, the active recovery was 4-6 min in intensity from 10 to 15 of scale of perceived exertion CR100.
  Arms: Interval Training
Other: Intermittent Training — The riders of intermittent training group completed 8 to 12 repetitions of 30 s all-out with 4 min of active recovery.
  Arms: Intermittent Training

SUMMARY:
The aerobic fitness is important for mountain bikers, but riders should also be able to generate maximal and supramaximal efforts in some crucial phases of the competition. Although there is an increase interest in high-intensity aerobic training, to investigators knowledge, there are no studies examining the effects of interval (INTV) or intermittent training (INTM) in mountain bikers. The aim of this study was to compare the effects of INTV and INTM on aerobic fitness variables (peak power output, Wmax, lactate threshold, and onset of blood lactate accumulation) but more importantly on performance as measured using a controlled mountain bike race, i.e. simulation. The investigators hypothesized that INTV and INTM training were equally effective in improving Wmax, Lactate threshold and onset of blood lactate accumulation, but INTV was superior in enhancing performance in mountai bike race simulation.This hypothesis is due to studies that have shown higher gains in performance with long duration of aerobic high intensity interval training in comparison to the shorter training at a higher intensity.

DETAILED DESCRIPTION:
The study is a controlled and randomized trial.

ELIGIBILITY:
Inclusion Criteria:

* Specific training in the mountain bike sport

Exclusion Criteria:

* Use of pharmacological substances

Ages: 20 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2010-10; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Interval Training and Performance in Mountain Bikers | Six weeks
  The aim of this study was to compare the effects of interval (INTV) and intermittent training (INTM) on aerobic fitness variables (peak power output, Wmax, lactate threshold, and onset of blood lactate accumulation) and performance as measured using a controlled MTB race, i.e. simulation. Pre to post differences were examined using two-way ANOVA, with a factor time on two levels (pre, post), and a factor group on two levels (INTV and INTM). Differences between groups post-training were also analyzed with ANCOVA using the pre-training values as covariate. These differences were calculated after log transforming the dependent variables. The difference between groups in the primary outcome (performance) was also analyzed using a magnitude-based inferences approach. The smallest worthwhile difference for the performance was considered to be 1%.

CONTACTS AND LOCATIONS:
Overall Officials: Tony M Santos, PhD, Principal Investigator — Gama Filho University
Locations (1):
- Gama Filho University, Rio de Janeiro, Rio de Janeiro, Brazil

REFERENCES:
- [Derived] Inoue A, Impellizzeri FM, Pires FO, Pompeu FA, Deslandes AC, Santos TM. Effects of Sprint versus High-Intensity Aerobic Interval Training on Cross-Country Mountain Biking Performance: A Randomized Controlled Trial. PLoS One. 2016 Jan 20;11(1):e0145298. doi: 10.1371/journal.pone.0145298. eCollection 2016. PMID 26789124